CLINICAL TRIAL: NCT05934227
Title: Long-term Effects of Sub Gingival Debridement Associated With Antibiotics in Individual Undergoing Maintenance Periodontal Therapy
Brief Title: Amoxicillin Plus Metronidazole in Periodontal Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Fernando O Costa, Titular Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5.957.583
Record Dates: First submitted 2023-06-17; First posted 2023-07-06 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Periodontitis; Periodontal Pocket
Keywords: amoxicillin; dental scaling; metronidazole; periodontal maintenance; periodontitis; root planing
MeSH Terms: conditions — Periodontitis; Periodontal Pocket | interventions — Amoxicillin

STUDY DESIGN:
Intervention Model Description: After clinical examination, participants will be randomly allocated into two treatment groups: 1) control group (SRP) - systemic administration of placebo after SRP (n = 25); 2) test group (SRP+AMX+MTZ) - systemic administration of AMX+MTZ after SRP (n=25).
Who Masked: Participant, Care Provider, Investigator
Masking Description: A random sequence will be generated (Excel, Microsoft Office 365) and participants will be allocated in the groups according to sequential numbered opaque envelopes. Each envelope containing one of the two treatments will be open only at the time of the periodontal procedure by the operator. Participants, as well as the researcher that evaluated treatment clinical outcomes won't know which group they were assigned.
  It will be ensure that the patient, the main researcher, the operator, the examiner and the statistician will be unaware of study groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): 1) scaling and root planing (SRP) plus systemic administration of placebo (n=25)
  Interventions: Other: placebo
- antibiotics (Experimental): 2) scaling and root planing (SRP) plus systemic administration of amoxicillin and metronidazole (n=25).
  Interventions: Drug: Amoxicillin 500 milligrams capsules plus metronidazole 400 milligrams

INTERVENTIONS:
Drug: Amoxicillin 500 milligrams capsules plus metronidazole 400 milligrams — supra and subgingival scaling and root planing (SRP) using manual and ultrasonic instruments in all residual pockets under anesthesia, performed within 2 consecutive days; systemic use of amoxicillin (500 milligrams) + metronidazole (400 milligrams) three times a day for 7 days after SRP
  Other Names: Amoxicillin Trihydrate; Amoxil
  Arms: antibiotics
Other: placebo — supra and subgingival scaling and root planing (SRP) using manual and ultrasonic instruments in all residual pockets under anesthesia, performed within 2 consecutive days; systemic use of placebo containing corn starch capsules three times a day for 7 days after SRP
  Arms: control

SUMMARY:
Gum disease require a lifetime supportive periodontal care aiming at preventing additional inflammation and bone resorption. During this phase it is also relevant to keep germs under acceptable levels through proper daily hygiene although patient's cooperation tends to decrease over time.

There are conflicting opinions regarding combination of dental scaling with antibiotics. This is why the present study was designed to evaluate the clinical and microbiological effects of combined therapy 1 year following supportive periodontal care. Fifty patients who voluntarily decide to participate will receive dental scaling associated with two different antibiotics or placebo capsules. Paper points will be used to collect dental plaque samples and levels of bacteria will be determined. Dental specialists will also perform clinical examinations. Patients would be available for 4 dental appointments: prior to and 3, 6 and 12 months after dental scaling.

DETAILED DESCRIPTION:
The benefits of amoxicillin (AMX) plus metronidazole (MTZ) adjunctive to scaling and root planing (SRP) require further investigation, particularly in individuals with a high occurrence of recurrent periodontal pockets under periodontal maintenance therapy (PMT). The aim of the study was to evaluate the clinical and microbiological outcomes of systemic AMX+MTZ adjunctive to SRP in patients with recurring sites [probing depth (PD) ≥5 mm) under PMT, after 1 year of follow-up, compared to SRP alone.

Methods: A randomized controlled clinical trial will be conducted with 50 individuals in a PMT program, which will be randomly allocate in two groups: control group (SRP and placebo; n=24) and test group (SRP and systemic MTZ+AMX; n=23). Participants of the present study will be selected from an open cohort study comprising individuals under a PMT program, who were monitored over 12 years of consecutive recall visits (from August 2009 to April 2023). Periodontal clinical parameters and subgingival biofilm samples will be collected by trained and calibrated examiners at baseline (T1), 3 (T2), 6 (T3) and 12 (T4) months after treatment. Microbiological analyses will be performed at T1, T2 and T4 by real-time quantitative polymerase chain reaction.

The percentage of residual pockets will be listed. Additionally, an overall mean PD value will be calculated for the treated sites initially measuring ≥ 5mm and clinical attachment loss (CAL) ≥ 3mm. Statistical testing for normality with respect to the distribution of study outcomes (clinical parameters) will be performed using the Kolmogorov-Smirnov test. Parametric and non-parametric tests (Chi-squared, Wilcoxon and Friedman tests) will be performed when appropriate. Spearman's correlation (r) will be used to evaluate the relationship between bacterial counts and periodontal condition between groups and evaluation times. All analyses will be performed using statistical software Statistical Package for the Social Sciences (SPSS) (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* individuals under a PMT program
* monitored over ~13 years of consecutive recall visits (from August 2009 to May 2023).
* individuals reclassified as stage III and IV periodontitis
* not having presented the following clinical endpoint in two consecutive PMT visits - presence of ≤4 sites with PD ≥5 mm
* non-diabetics
* non-smokers
* no antibiotic use for any purpose within 3 months prior to entering the study

Exclusion Criteria:

* pregnant or lactating women
* smokers
* presence of systemic diseases that could affect the progression of periodontitis long-term administration of anti-inflammatory drugs,
* need for antibiotic premedication for routine dental therapy and
* allergy to metronidazole or amoxicillin

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
whole-mouth periodontal pocket depth improvement | baseline and 12 months
  mean pocket depth (PD) in millimeters
changes in percentage of deep periodontal pocket | baseline and 12 months
  proportion of sites with PD ≥5 millimeters

SECONDARY OUTCOMES:
total bacterial load in sub gingival samples | baseline and 3 months
  mean total bacterial load
levels of target species in sub gingival samples | baseline and 3 months
  mean levels of periodontal pathogens

CONTACTS AND LOCATIONS:
Overall Officials: Fernando O Costa, PhD, Principal Investigator — Titular Professor in periodontics
Locations (1):
- Federal University of Minas Gerais, Dental School, Belo Horizonte, Minas Gerais, Brazil